CLINICAL TRIAL: NCT03168854
Title: A Phase 1, Two Arm, Open Label Trial to Evaluate the Safety, Immunogenicity and Preliminary Efficacy of Genetically-attenuated p52-/p36-/sap1- Plasmodium Falciparum Parasites (GAP3KO) Administered Via the Bite of Infected Anopheles Stephensi Mosquitoes to Malaria-Naïve Adults Living in the United States
Brief Title: Trial to Evaluate the Safety, Immunogenicity and Protective Efficacy of Three or Five Administrations of GAP3KO Sporozoites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-0088
Record Dates: First submitted 2017-05-18; First posted 2017-05-30 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2017-12-11

CONDITIONS: Plasmodium Falciparum Infection
Keywords: Anopheles stephensi Mosquitoes; GAP3KO; Genetically-attenuated; Malaria-Naïve Adults; Phase 1; Plasmodium falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- GAP Arm 1 (Experimental): 10 subjects will receive 5 vaccinations: the GAP3KO vaccine administered by the bite of approximately 200 infected A. Stephensi mosquitoes at weeks 0, 4, 8, 12, and 20 for a maximum cumulative dose of 1000 GAP3KO bites per subject
  Interventions: Biological: Genetically-attenuated p52-/p36-/sap1- Plasmodium falciparum parasite (GAP3KO) strain; Other: Malaria challenge
- GAP Arm 2 (Experimental): 6 subjects will receive 3 vaccinations: the GAP3KO vaccine administered by the bite of approximately 200 infected A. Stephensi mosquitoes at weeks 8, 12, and 20 for a maximum cumulative dose of 600 GAP3KO bites per subject
  Interventions: Biological: Genetically-attenuated p52-/p36-/sap1- Plasmodium falciparum parasite (GAP3KO) strain; Other: Malaria challenge
- Malaria-naive Infectivity Control Arm (Active Comparator): 6 healthy volunteers will receive challenge with wild type Plasmodium falciparum NF54 sporozoites through the bites of five infectious A. stephensi moquitoes using standard CHMI procedures
  Interventions: Other: Malaria challenge

INTERVENTIONS:
Biological: Genetically-attenuated p52-/p36-/sap1- Plasmodium falciparum parasite (GAP3KO) strain — Genetically attenuated parasite created by triple deletion (GAP3KO) by deleting the P52, P36, and SAP1 genes in the NF54 wild-type (WT) strain of Plasmodium falciparum (Pf p52(-)/p36(-)/sap1(-) GAP).
  Arms: GAP Arm 1; GAP Arm 2
Other: Malaria challenge — Exposure to mosquitoes infected with P. falciparum.

SUMMARY:
This Phase 1 trial will include 16 subjects who will receive the Genetically-attenuated p52-/p36-/sap1- Plasmodium falciparum Parasites (GAP3KO) vaccine administered by the bite of approximately 200 infected Anopheles stephensi Mosquitoes in a controlled clinical environment and 12 Controlled Human Malaria Infection (CHMI) infectivity controls (six for each of the two CHMIs). Subjects will be observed for adverse events after each GAP3KO administration. Solicited local and systemic Adverse Events (AEs) will be recorded on a memory aid beginning of the day of first vaccine administration and continuing through 28 days after the last administration. During the vaccination phase clinical laboratory evaluations for safety will be performed on venous blood. Unsolicited AEs will be collected from the day of first vaccination through 28 days after last vaccination and serious adverse events (SAEs) will be collected from the day of first GAP3KO administration through the end of study follow-up. Subjects will be monitored for possible breakthrough peripheral parasitemia with qRT-PCR testing. Four weeks after the last GAP3KO administration, all subjects who completed the immunization phase (up to 16) and a group of six malaria-naïve infectivity controls will be challenged on the same day with wild-type Plasmodium falciparum NF54 sporozoites. Approximately twenty-six weeks after that challenge, all of the protected subjects in Arms 1 and 2 (up to 16) and another six malaria-naïve infectivity controls will receive five infectious A. stephensi mosquito bites on the same day using standard CHMI procedures. For subjects in Study Arms 1 and 2 without documented parasitemia additional post-CHMI follow-ups will occur. For subjects in Study Arms 1 and 2 with documented parasitemia after the first CHMI or who are discontinued for other reasons after the first CHMI, and for the infectivity controls, additional follow ups will occur. Serious Adverse Events (SAEs) will be recorded from the day of CHMI through the end of study follow up and clinical laboratory evaluations for safety will be performed on Day 29 and as clinically indicated (all subjects) and, for subjects with documented parasitemia, on the day malaria treatment is initiated and three days after malaria treatment is initiated. The primary objectives are: 1) To assess the safety and reactogenicity of candidate GAP3KO malaria vaccine when administered by the bite of approximately 200 infected mosquitoes on a five dose schedule, with the first four vaccinations given four weeks apart and the fifth vaccination given eight weeks after the fourth vaccination, and on a three dose schedule, with the second vaccination given four weeks after the first vaccination and the third vaccination given eight weeks after the second vaccination, to healthy malaria-naïve adults aged 18 through 50 years , 2) To confirm attenuation of GAP3KO parasites by assessing the occurrence of breakthrough peripheral parasitemia from the time of first GAP3KO administration through 28 days after last GAP3KO administration.

DETAILED DESCRIPTION:
This Phase 1 trial will include 16 subjects in Study Arms 1 and 2 who will receive the Genetically-attenuated p52-/p36-/sap1- Plasmodium falciparum Parasites (GAP3KO) vaccine administered by the bite of approximately 200 infected Anopheles stephensi Mosquitoes in a controlled clinical environment and 12 Controlled Human Malaria Infection (CHMI) infectivity controls (six for each of the two CHMIs). Subjects will be observed for adverse events for at least 60 minutes after each GAP3KO administration. Solicited local and systemic Adverse Events (AEs) will be recorded on a memory aid beginning of the day of first vaccine administration and continuing through 28 days after the last administration. During the vaccination phase clinical laboratory evaluations for safety will be performed on venous blood. Unsolicited AEs will be collected from the day of first vaccination through 28 days after last vaccination and serious adverse events (SAEs) will be collected from the day of first GAP3KO administration through the end of study follow-up. Subjects will be monitored for possible breakthrough peripheral parasitemia with qRT-PCR testing. Four weeks after the last GAP3KO administration, all subjects who completed the immunization phase (up to 16) and a group of six malaria-naïve infectivity controls will be challenged on the same day with wild-type Plasmodium falciparum NF54 sporozoites. Approximately twenty-six weeks (six months) after that challenge, all of the protected subjects in Arms 1 and 2 (up to 16) and another six malaria-naïve infectivity controls will receive five infectious A. stephensi mosquito bites on the same day using standard CHMI procedures. For subjects in Study Arms 1 and 2 without documented parasitemia additional post-CHMI follow-ups will occur. For subjects in Study Arms 1 and 2 with documented parasitemia after the first CHMI or who are discontinued for other reasons after the first CHMI, and for the infectivity controls, additional follow ups will occur. Serious Adverse Events (SAEs) will be recorded from the day of CHMI through the end of study follow up and clinical laboratory evaluations for safety will be performed on Day 29 and as clinically indicated (all subjects) and, for subjects with documented parasitemia, on the day malaria treatment is initiated and three days after malaria treatment is initiated. The primary objectives are: 1) To assess the safety and reactogenicity of candidate GAP3KO malaria vaccine when administered by the bite of approximately 200 infected mosquitoes on a five dose schedule, with the first four vaccinations given four weeks apart and the fifth vaccination given eight weeks after the fourth vaccination, and on a three dose schedule, with the second vaccination given four weeks after the first vaccination and the third vaccination given eight weeks after the second vaccination, to healthy malaria-naïve adults aged 18 through 50 years , 2) To confirm attenuation of GAP3KO parasites by assessing the occurrence of breakthrough peripheral parasitemia from the time of first GAP3KO administration through 28 days after last GAP3KO administration. The secondary objectives are: 1) To assess the efficacy of GAP3KO vaccine given on a five dose schedule and GAP3KO vaccine given on a three dose schedule against malaria challenge four weeks after last vaccination, and re-challenge 26 weeks (six months) after the first challenge, using standard controlled human malaria infection (CHMI) procedures, 2) To assess humoral and cell-mediated immune responses to malaria antigens induced by GAP3KO administration and by CHMI.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in this study.

1. 18 through 50 years of age, inclusive.
2. Able and willing to participate for the duration of the study and able to understand and comply with planned study procedures.
3. Able and willing to provide written (not proxy) informed consent.
4. Provides informed consent before initiation of any study procedure, correctly answers = / > 80 percent of questions* on the post consent quiz and is available for all study visits.

   *Subjects who score less than 80 percent may retake the quiz one time and are excluded if the second test is also less than 80 percent.
5. Is in good health, as judged by the investigator, and determined by medical history and physical examination.

   *Existing medical diagnoses or conditions (except those in the Subject Exclusion Criteria) must be deemed as stable. A stable medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last three months (90 days) and health outcomes of the specific disease are considered to be within acceptable limits in the last six months (180 days). Any change due to change of health care provider, insurance company, or that is done for financial reasons, as long as in the same class of medication, will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a violation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of solicited events and immunogenicity.
6. Women of childbearing potential* must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to each mosquito exposure**.

   * Not sterilized via bilateral tubal ligation, bilateral oophorectomy, or hysterectomy, or, if menopausal, still menstruating or < 1 year of the last menses.

     * Study vaccination or CHMI
7. Women of childbearing potential must have used a highly effective form of contraception* in the 30 days prior to their first mosquito exposure**.

   *Highly effective single forms of contraception include abstinence from sexual activity that could lead to pregnancy, monogamous relationship with vasectomized partner who has been vasectomized for six months or more prior to enrollment, successful Essure (R) placement (permanent, non-surgical, non-hormonal sterilization) with documented confirmation test at least three months after the procedure, or use of effective intrauterine devices or the contraceptive implant (Nexplanon). If none of the highly effective single forms of contraception is used, a combination of an acceptable barrier method and an acceptable hormonal method must be used. Acceptable barrier methods include condom (male or female) and a spermicide (cream, film, foam, or gel), diaphragm or cervical cap with spermicide, and the birth control sponge. Acceptable hormonal methods include birth control patch, shot (Depo-Provera), and pills, and the vaginal ring (NuvaRing).

   **Study vaccination or CHMI.
8. Women of childbearing potential must agree to continue use of a highly effective form of contraception through 90 days after their last mosquito exposure.
9. For women, must not be breastfeeding or plan to start breastfeeding at any time before the end of study follow up.
10. At low (< / = 10 percent) 5-year cardiovascular risk*. *Per the risk prediction method of Gaziano (https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2864150/). Risk for persons < 35 years of age will be based on the age 35-44 group.
11. No history of malaria infection or vaccination, residence in a malaria-endemic area for > / = 5 years, or participation in a malaria research study*.

    *Participation without exposure to malaria infection or to a malaria vaccine is not exclusionary.
12. No receipt of malaria prophylaxis or travel to a malaria-endemic area in the six months prior to first mosquito exposure.
13. No receipt of blood products or immunoglobulin within six months prior to, or donation of a unit of blood within two months prior to, enrollment.
14. Weight > / = 50 kg and body mass index (BMI) < 35 kg/m^2.
15. Negative serology for HIV 1/2*.

    *If the ELISA is positive, HIV confirmation should be performed. If the HIV Western Blot is not consistent with HIV infection, the subject may be enrolled. A past subject in an HIV vaccine trial who has a positive antibody ELISA may participate if the Western Blot is not consistent with pending seroconversion or positive or an HIV PCR assay result is below the level of detection of HIV.
16. Negative hepatitis B surface antigen and hepatitis C virus antibody.
17. No Grade 1 or higher screening clinical lab value*.

    *Screening clinical labs include blood tests (white blood count [WBC], hemoglobin, platelet count, creatinine, and alanine aminotransferase [ALT]) and urine dipstick tests (protein and hemoglobin). Any Grade 1 or higher value for any screening test will exclude the subject from enrollment with the exception of hematuria > / = 1 + detected concurrent with endometrial bleeding for females. In this situation, the test can be repeated if clinically warranted but is not considered an indicator of poor health status or increased risk and so is not a contraindication to enrollment.
18. Screening ECG with no clinically significant abnormalities*.

    *Pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial or ventricular contractions; right or left bundle branch block; QT / QTc interval > 450 ms; or advanced (secondary or tertiary) A-V heart block.
19. No known allergy to mosquito bites, chloroquine, hydroxychloroquine, amodiaquine atovaquone, proguanil, non-steroidal anti-inflammatory drugs, or acetaminophen.
20. No known sickle cell trait or other hemoglobinopathy.
21. Negative sickle cell screening laboratory test.
22. Does not plan to undergo surgery (elective or otherwise) between screening and the end of the study.
23. No dermatologic abnormalities in either forearm that could impair assessment of local reactions.
24. No history of psoriasis or porphyria.
25. No history of G6PD deficiency.
26. No contraindication to repeated phlebotomy*. *Such as minimal venous access or recent history of anemia.
27. Reachable (24/7) by mobile phone during the duration of the study period and willing to provide two close contacts to assist with making contact.
28. Lives in the greater Seattle area and within an approximately one hour commute to the study research clinic.
29. Willing to avoid non-study related blood donation for the duration required by the blood bank* following last mosquito exposure.

    *Bloodworks Northwest prohibits donation from persons who have had malaria.
30. Agrees not to travel to a malaria endemic region during the entire course of the trial.
31. Agrees not to travel away from the greater Seattle area in the 14 days after a study immunization*, and from the day of CHMI until the end of malaria treatment visits.

    * Subjects in Study Arms 1 and 2.

Exclusion Criteria:

A subject meeting any of the following exclusion criteria are not eligible for enrollment.

1. Use of any antibiotic or drug with antimalarial properties within 28 days prior to first mosquito exposure or planned use during the study period.
2. Any clinically significant acute or chronic medical condition* or need for chronic medications** that, in the opinion of the investigator, will interfere with immunity or affect safety.

   *Includes, but is not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions.

   **Receipt of systemic, prescription medications for the treatment of chronic medical conditions or variations of normal physiologic functions are permissible if, in the opinion of the investigator, they are used for conditions that are not clinically significant and would not impact the effectiveness of the vaccine or the safety of the subject or the safety and immunogenicity outcomes of the protocol. Use of systemic, over-the-counter medications and PRN systemic, prescription medications are allowed if, in the opinion of the investigator, they pose no additional risk to subject safety, vaccine efficacy or assessment of immunogenicity/reactogenicity. Topical (except corticosteroid) medications, nasal (including corticosteroid) medications, vitamins, and supplements are permissible. Following enrollment, use of topical corticosteroid medications for treatment of GAP3KO administration reactions is permissible. Any drug with antimalarial properties is not permissible.
3. Asthma, other than mild, well-controlled asthma*.

   *Cold or exercise-induced asthma controlled with inhaled medications other than inhaled corticosteroids is permissible. Subjects should be excluded if they require daily bronchodilator use, or have had an asthma exacerbation requiring oral/parenteral steroid use or have used theophylline or inhaled corticosteroids in the past year
4. Known atherosclerotic cardiovascular disease or history of myocardial infarction, pericarditis, or myocarditis.
5. Diabetes mellitus.
6. History of a psychiatric condition that may make study compliance difficult, such as schizophrenia or bipolar disorder*.

   *Includes persons with psychoses or history of suicide attempt or gesture in the 3 years before study entry or an ongoing risk for suicide.
7. Chronic or active neurologic condition (including seizures and migraine headaches).
8. Autoimmune disease (autoimmune thyroid disease is permissible and vitiligo or mild eczema not requiring chronic therapy is permissible).
9. Known or suspected congenital or acquired immunodeficiency including anatomic or functional asplenia* or immunosuppression as a result of underlying illness or treatment.

   *Any splenectomy is exclusionary.
10. Abuse of alcohol or drugs that, in the opinion of the investigator, may interfere with ability to comply with the protocol or increase risk to subject's health during the study period.
11. Active neoplastic disease*.

    *Subjects with a history of malignancy may be included if treated by surgical excision or if treated by chemotherapy or radiation therapy and has been observed for a period that in the investigator's estimation provides a reasonable assurance of sustained cure (not less than 36 months). Cervical neoplasia under surveillance is acceptable.
12. Chronic topical or systemic corticosteroid use*.

    *Corticosteroid nasal sprays for allergic rhinitis are permissible. Persons using a topical corticosteroid for a limited duration for mild uncomplicated dermatitis such as poison ivy or contact dermatitis prior to enrollment may be enrolled the day after their therapy is completed. Oral or parenteral (intravenous, intramuscular, subcutaneous) corticosteroids given for non-chronic conditions not expected to recur are permissible if, within the year prior to enrollment, the longest course of therapy was no more than 14 days and no oral or parenteral corticosteroids were given within 30 days prior to enrollment. Intraarticular, bursal, tendon, or epidural injections of corticosteroids are permissible if the most recent injection was at least 30 days prior to enrollment. Topical or systemic corticosteroid use for study related adverse events is not exclusionary.
13. Receipt or planned receipt of inactivated vaccine or allergy desensitization injection within 14 days before or after a mosquito exposure.
14. Receipt or planned receipt of live attenuated vaccine within 28 days before or after a mosquito exposure.
15. Current use of tenofovir/emtricitabine (Truvada).
16. Receipt of any experimental agent* within 30 days prior to screening or planned receipt prior to the end of the study.

    *Vaccine, drug, biologic, device, blood product, or medication.
17. Plans to enroll in another clinical trial* that could interfere with safety assessment of the investigational product at any time during the study period.

    *Includes trials that have a study intervention such as a drug, biologic, or device.
18. Systolic blood pressure > / = 161 mm Hg or diastolic blood pressure > / = 96 mm Hg.
19. Resting heart rate < / = 49 or > / = 101 beats per minute.
20. Oral temperature > / = 38 degree Celsius (100.4 degree Fahrenheit).
21. Acute febrile illness (oral temperature = / > 38 degree Celsius [100.4 degree Fahrenheit]) or other acute illness within three days prior to mosquito exposure*.

    *Note for afebrile, acute illness only: If a subject is afebrile, his/her acute illness is nearly resolved with only minor residual symptoms remaining, and, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol, the subject may receive the subsequent study vaccination or CHMI without further approval from the DMID Medical Officer.
22. Is using or intends to use within 28 days after a mosquito exposure a medication with a known interaction with atovaquone-proguanil* or chloroquine**.

    *Includes, for example, tetracycline (may reduce atovaquone concentrations), or metoclopramide (may reduce bioavailability of atovaquone).

    **Includes, for example, cimetidine, metoclopramide, carbamazepine, phenytoin, St. John's wort, and antidepressants. Antacids and kaolin may reduce absorption of chloroquine but can be administered if separated by at least 4 hours from intake of chloroquine.
23. Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Breakthrough peripheral parasitemia defined as two positive qRT-PCR assays with parasite densities of > /= 20 estimated parasites/mL from blood samples obtained at least six hours apart or a positive TBS | First GAP3KO administration through 28 days after last GAP3KO administration
Laboratory toxicities related to vaccination that are classified as Grade 3(Severe). Grade 3 being defined as events that interrupt the subject's usual daily activities and may require systemic drug therapy or other treatment. | First GAP3KO administration through 14 days after last GAP3KO administration
Serious adverse events (SAEs) considered related to vaccination | First GAP3KO administration through the end of study follow-up, up to 20 months after first study visit.
Solicited local adverse events (AEs) | First GAP3KO administration through 28 days after last GAP3KO administration
Solicited systemic adverse events (AEs) | First GAP3KO administration through 28 days after last GAP3KO administration
Unsolicited AEs considered related to vaccination | First GAP3KO administration through 28 days after last GAP3KO administration

SECONDARY OUTCOMES:
Documented malaria infection, defined as a positive qRT-PCR assays with parasite densities of > /= 20 estimated parasites/mL, from blood samples obtained at least six hours apart or a positive TBS | 28 days following CHMI
Frequencies of PBMCs and PBMC subsets secreting specific cytokines on stimulation with whole sporozoites and potentially specific malaria antigens by intracellular cytokine staining (ICS) of cells | Pre-vax visit, Pre-CHMI visit
Levels of IgG antibodies to circumsporozoite protein (CSP) measured by ELISA on serum samples | Pre-vax visit, Pre-CHMI visit

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States